CLINICAL TRIAL: NCT05389410
Title: Comparison of Surgical Wound Healing and Complications Following Revision Hip and Knee Replacements, Utilising a 7-day Versus 14-day Negative Pressure Wound Therapy (NPWT) Dressing. A Randomised Controlled Trial.
Brief Title: PICO 7 vs PICO 14 in Revision Hip and Revision Knee Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RL1 786
Record Dates: First submitted 2022-05-16; First posted 2022-05-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Surgical Wound
Keywords: Revision hip and revision knee surgery
MeSH Terms: conditions — Surgical Wound | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revision Hip surgery (Experimental): Participants will be randomised to PICO 7 or PICO 14 intervention.
  Interventions: Device: PICO 7; Device: PICO 14
- Revision knee surgery (Active Comparator): Participants will be randomised to PICO 7 or PICO 14 intervention.
  Interventions: Device: PICO 7; Device: PICO 14

INTERVENTIONS:
Device: PICO 7 — Participant will receive 7 days of NPWT following revision hip or revision knee surgery.
  Other Names: 7 day NPWT
Device: PICO 14 — Participant will receive 14 days of NPWT following revision hip or revision knee surgery.
  Other Names: 14 day NPWT

SUMMARY:
This is a single-site trial, and it has been designed to compare a revision hip cohort with a revision knee cohort. All consecutive eligible patients, under the care of participating Co-Investigator Orthopaedic Surgeons, are approached for recruitment into the study.

Eligible patients wishing to participate must require either revision hip or revision knee surgery and consent to be randomised to either NPWT PICO dressing for 7-day therapy (PICO 7) or NPWT PICO 14-day therapy (PICO 14).

82 Revision Hips and 82 Revision Knee participants, with 41* of each cohort randomised to either a 7-day or a 14-day NPWT dressing treatment duration period. The 7-day cohort will be treated with PICO7 dressings and pumps, and the 14-day cohort will be treated with PICO14 dressings.

*Randomisation will be stratified, so it will continue until there are at least 41 participants in each cohort.

DETAILED DESCRIPTION:
Although the efficacy of these dressings is well established in promoting wound healing, the duration of application particularly in revision surgeries, where the surgery has been carried out though old scar tissues is however undetermined at present. The few published studies regarding this do show a benefit, however, they do not address the potential issues surrounding late wound breakdown and the duration of the NPWT on the wound 4,5.

Therefore a proposed randomised study to evaluate whether one-week of negative pressure wound therapy is sufficient or whether a two-week therapy duration is warranted.

This will be done by randomising a minimum of 82 patients who are scheduled for revision hip surgery and 82 patients who are scheduled for revision knee surgery into either a "control group" or a "study group".

The 'control group' cohort will receive a NPWT PICO 7 dressing and pump for a period of week, followed by a hydrocolloid dressing or other standard dressing applied thereafter. The 'study group' cohort will receive a NPWT PICO 14 dressing and pump for a period of 2 weeks, with a dressing change at one week. The pump will be paused during the dressing change, restarting it again once the new dressing has been applied and sealed for another week's NPWT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be over the age of 18 years.
* Participants undergoing aseptic revision hip or aseptic revision knee surgery procedure (a single stage revision procedure).
* Participants must be willing and be able to make all the required study visits to be seen by the research team at the Outpatients department at RJAH.
* Participants must be able to follow instructions.

Exclusion Criteria:

* Revisions for infection, where the nature of the infection has a significant influence on the wound healing, discharge, and length of stay.
* Subjects with a history of poor compliance with medical treatment.
* Subjects with contraindications (as per the PICO Instructions for use) or hypersensitivity to the use of the NPWT PICO dressing product or its components e.g.: silicone adhesives, polyurethane films, acrylic adhesives, polyethylene fabrics and super- absorbent powders (polyacrylates) contained within the dressing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
The extent of wound exudate graded 1-4. This is measured by the extent of staining on the dressing at 1-week post-surgery (both study and control groups) and 2 weeks post-surgery (study group only). | Within the first 2 weeks post-surgery
  The extent of wound exudate graded 1-4 (measured by the extent of staining on the dressing) at 1 week and 2 weeks at follow up appointments.
  Grading of wound exudate levels and the amount of exudate on the coverage of the dressing:
  Grade 0 None No staining Grade 1 Light < 25% Grade 2 Moderate 25% to 50% Grade 3 Heavy 50% to 75% Grade 4 Overt > 75%
Late wound dehiscence or wound discharge (discharge from the wound once the PICO dressing has been discontinued). | For the study duration, up to 6 weeks post-surgery.
  If there is any wound discharge after the PICO has been discontinued as per the protocol.
  The duration of wound discharge (any patients experiencing persistent discharge beyond 48 hrs will be brought back to clinic and dealt appropriately as per the Consultants preferred management methods).
  If there is any wound dehiscence or breakdown (patients will be brought back to clinic and again, dealt appropriately as per consultants preferred wound management method).
  The management of persistent wound discharge may require hospitalisation, wound washout or continued and/or prolonged use of a PICO dressing. These are all part of the standard of care at RJAH, but their use does vary slightly, depending on individual preferences of the supervising Surgeon.
Observance of the formation of wound complications, specifically superficial wound infection, and deep wound infection. | For the study duration, up to 6 weeks post-surgery.
  The number of wound complications, specifically concerning superficial wound infections and deep wound infections. The patient will be monitored at 1 week (clinic visit), 2 week (clinic visit), 3 week (phone call), and 6 weeks (clinic visit).

SECONDARY OUTCOMES:
Wound appearance documented by photographs from before the dressing is applied in theatre to 6 weeks post-surgery follow up visit. | For the study duration, up to 6 weeks post-surgery.
  The appearance of the wound at the 1-week clinic visit, where the dressing is changed or PICO therapy discontinued, depending on the treatment arm that the patient has been randomised to, the 2-week clinic visit, where the "study" cohort of patients will have their second dressing removed and at the 6-week clinic visit. The evidence of the wound appearance at these time points will be documented through photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Sudheer L Karlakki, Principal Investigator — The Robert Jones and Agnes Hunt Orthopaedic Hospital Foundation Trust
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Malmsjo M, Huddleston E, Martin R. Biological effects of a disposable, canisterless negative pressure wound therapy system. Eplasty. 2014 Apr 2;14:e15. eCollection 2014. PMID 24741386
- [Result] Nherera LM, Trueman P, Karlakki SL. Cost-effectiveness analysis of single-use negative pressure wound therapy dressings (sNPWT) to reduce surgical site complications (SSC) in routine primary hip and knee replacements. Wound Repair Regen. 2017 May;25(3):474-482. doi: 10.1111/wrr.12530. Epub 2017 May 3. PMID 28370637
- [Result] Helito CP, Bueno DK, Giglio PN, Bonadio MB, Pecora JR, Demange MK. NEGATIVE-PRESSURE WOUND THERAPY IN THE TREATMENT OF COMPLEX INJURIES AFTER TOTAL KNEE ARTHROPLASTY. Acta Ortop Bras. 2017 Mar-Apr;25(2):85-88. doi: 10.1590/1413-785220172502169053. PMID 28642657
- [Result] Miyahara HS, Serzedello FR, Ejnisman L, Lima ALLM, Vicente JRN, Helito CP. INCISIONAL NEGATIVE-PRESSURE WOUND THERAPY IN REVISION TOTAL HIP ARTHROPLASTY DUE TO INFECTION. Acta Ortop Bras. 2018;26(5):300-304. doi: 10.1590/1413-785220182605196038. PMID 30464709
- [Result] Newman JM, Siqueira MBP, Klika AK, Molloy RM, Barsoum WK, Higuera CA. Use of Closed Incisional Negative Pressure Wound Therapy After Revision Total Hip and Knee Arthroplasty in Patients at High Risk for Infection: A Prospective, Randomized Clinical Trial. J Arthroplasty. 2019 Mar;34(3):554-559.e1. doi: 10.1016/j.arth.2018.11.017. Epub 2018 Nov 17. PMID 30545653
- [Result] Karlakki SL, Hamad AK, Whittall C, Graham NM, Banerjee RD, Kuiper JH. Incisional negative pressure wound therapy dressings (iNPWTd) in routine primary hip and knee arthroplasties: A randomised controlled trial. Bone Joint Res. 2016 Aug;5(8):328-37. doi: 10.1302/2046-3758.58.BJR-2016-0022.R1. PMID 27496913
- [Result] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Result] Barbachano Y, Coad DS. Inference following designs which adjust for imbalances in prognostic factors. Clin Trials. 2013 Aug;10(4):540-51. doi: 10.1177/1740774513493367. Epub 2013 Jul 5. PMID 23832671
- [Result] The ASA's Statement on p-values: Context, Process, and Purpose
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343